CLINICAL TRIAL: NCT01592045
Title: A Comparative Pharmacokinetic and Safety Study of Chimeric Monoclonal Antibody ch14.18 With Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF), Interleukin-2 (IL-2) and Isotretinoin in High Risk Neuroblastoma Patients Following Myeloablative Therapy
Brief Title: ch14.18 Pharmacokinetic Study in High-risk Neuroblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIV-NB-201
Record Dates: First submitted 2012-04-30; First posted 2012-05-04 (Estimated); Results first posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-08

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab; Granulocyte-Macrophage Colony-Stimulating Factor; aldesleukin; Interleukin-2; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence 1 (Experimental): UTC ch14.18 for two courses and NCI ch14.18 for three courses
  Interventions: Biological: ch14.18 -NCI; Biological: ch14.18-UTC; Biological: Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF); Biological: Aldesleukin (IL-2); Drug: Isotretinoin
- Sequence 2 (Experimental): NCI ch14.18 for two courses and UTC ch14.18 for three courses
  Interventions: Biological: ch14.18 -NCI; Biological: ch14.18-UTC; Biological: Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF); Biological: Aldesleukin (IL-2); Drug: Isotretinoin

INTERVENTIONS:
Biological: ch14.18 -NCI — 25 mg/m^2/day IV for four consecutive days
Biological: ch14.18-UTC — 17.5 mg/m^2/day IV for four consecutive days
Biological: Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) — GM-CSF will be administered SC at a dose of 250 mcg/m^2/day for 14 days during Courses 1, 3, and 5.
Biological: Aldesleukin (IL-2) — Aldesleukin (IL-2) will be administered IV at a dose of 3 MIU/m^2/day for the first week and at a dose of 4.5 MIU/m^2/day for the second week during Courses 2 and 4.
Drug: Isotretinoin — Isotretinoin (13-cis-retinoic acid; ISOT) will be administered by mouth over six courses as follows:
  If weight > 12 kg: 80 mg/m^2/dose twice daily (total daily dose is 160 mg/m^2/day, divided twice daily).
  If weight ≤ 12 kg: 2.67 mg/kg/dose twice daily (total daily dose is 5.33 mg/kg/day, divided twice daily).
  Other Names: 13-cis-retinoic acid

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (blood levels) and safety of chimeric (ch) 14.18 manufactured by two independent drug makers (United Therapeutics [UTC] or the National Cancer Institute [NCI]).

DETAILED DESCRIPTION:
This is a multi-center, randomized, open-label, two-sequence, cross-over study for eligible subjects with high-risk neuroblastoma to assess the comparability of ch14.18 manufactured with UTC drug product and ch14.18 manufactured with NCI drug product. Subjects will be randomly allocated to receive ch14.18 manufactured by UTC or NCI during Courses 1 and 2 followed by ch14.18 manufactured by other manufacturer (UTC or NCI) during Courses 3, 4, and 5.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high-risk neuroblastoma
* 8 years of age or younger at diagnosis of high-risk neuroblastoma
* Patients must have completed therapy including intensive induction followed by autologous stem cell transplantation (ASCT) and radiotherapy

  * Radiotherapy may be waived for patients who either have small adrenal masses which are completely resected up front, or who never have an identifiable primary tumor
* Must meet the International Neuroblastoma Response Criteria (INRC) for CR, VGPR, or PR for primary site, soft tissue metastases, and bone metastases AND must also meet the protocol specified criteria for bone marrow response as follows:

  * No more than 10% tumor (of total nucleated cellular content) seen on any specimen from a bilateral bone marrow aspirate/biopsy
* Patient who have no tumor seen on the prior bone marrow, and then have ≤ 10% tumor on any of the bilateral marrow aspirate/biopsy specimens done at pre-ASCT and/or pre-enrollment evaluation will also be eligible
* No more than 12 months from starting the first induction chemotherapy after diagnosis to the date of ASCT

  * For patients who became high-risk neuroblastoma after initial non-high risk disease, the 12 months period should start from the date of induction therapy for high-risk neuroblastoma to the date of ASCT
* No progressive disease at time of registration except for protocol-specified bone marrow response
* Adequate hematological, renal, hepatic, pulmonary and cardiac function
* CNS toxicity < Grade 2

Exclusion Criteria:

* Prior anti-GD2 antibody therapy
* Prior vaccine therapy for neuroblastoma
* Concurrent anti-cancer or immunosuppressive therapy

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Araz Marachelian, MD, Study Chair — Children's Hospital Los Angeles
Locations (13):
- United States (13):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Children's Mercy Hospital (Kansas), Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: UTC ch14.18 for two courses followed by NCI ch14.18 for three courses
  ch14.18 -NCI: 25 mg/m^2/day IV for four consecutive days
  ch14.18-UTC: 17.5 mg/m^2/day IV for four consecutive days
  Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF): GM-CSF will be administered SC at a dose of 250 mcg/m^2/day for 14 days during Courses 1, 3, and 5.
  Aldesleukin (IL-2): Aldesleukin (IL-2) will be administered IV at a dose of 3 MIU/m^2/day for the first week and at a dose of 4.5 MIU/m^2/day for the second week during Courses 2 and 4.
  Isotretinoin: Isotretinoin (13-cis-retinoic acid; ISOT) will be administered by mouth over six courses as follows:
  If weight > 12 kg: 80 mg/m^2/dose twice daily (total daily dose is 160 mg/m^2/day, divided twice daily).
  If weight ≤ 12 kg: 2.67 mg/kg/dose twice daily (total daily dose is 5.33 mg/kg/day, divided twice daily).
- Sequence 2: NCI ch14.18 for two courses followed by UTC ch14.18 for three courses
  ch14.18 -NCI: 25 mg/m^2/day IV for four consecutive days
  ch14.18-UTC: 17.5 mg/m^2/day IV for four consecutive days
  Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF): GM-CSF will be administered SC at a dose of 250 mcg/m^2/day for 14 days during Courses 1, 3, and 5.
  Aldesleukin (IL-2): Aldesleukin (IL-2) will be administered IV at a dose of 3 MIU/m^2/day for the first week and at a dose of 4.5 MIU/m^2/day for the second week during Courses 2 and 4.
  Isotretinoin: Isotretinoin (13-cis-retinoic acid; ISOT) will be administered by mouth over six courses as follows:
  If weight > 12 kg: 80 mg/m^2/dose twice daily (total daily dose is 160 mg/m^2/day, divided twice daily).
  If weight ≤ 12 kg: 2.67 mg/kg/dose twice daily (total daily dose is 5.33 mg/kg/day, divided twice daily).
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2
Started | 14 | 14
Completed Course 1 | 13 | 14
Completed Course 2 | 13 | 13
Completed Course 3 | 11 | 13
Completed Course 4 | 11 | 12
Completed Course 5 | 9 | 12
Completed | 9 | 12
Not Completed | 5 | 2
Not completed — Disease Progression | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Moved out of country | 2 | 0

BASELINE CHARACTERISTICS:
Population: Twenty-eight subjects were enrolled in this study with all subjects receiving at least one dose of study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Full Range); unit: years] | 4 [2 to 7] | 4 [1 to 9] | 4 [1 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Pre-ASCT Response [Number; unit: participants] — At pre-ASCT evaluation, subjects must have met the International Neuroblastoma Response Criteria (INRC) for complete response (CR), very good partial response (VGPR) or partial response (PR) for primary site, soft tissue metastases, and bone metastases. Subjects who met those criteria were also required to meet the protocol specified criteria for bone marrow response.
  participants
    Complete Response (CR) | 5 | 3 | 8
    Very Good Partial Response (VGPR) | 5 | 4 | 9
    Partial Response (PR) | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Curve (AUC)
Description: Twenty-two PK samples will be obtained at the following timepoints:
  Courses 1 and 3:
  Day: 0 Days: 3, 4, 5 and 6: post ch14.18 Days 7:10 to 14 hours post ch14.18 Days 9 to 11: Single sample Days 14 to 17: Single sample
  Courses 2 and 4:
  Day 0: Pre-IL-2 Day 7: Pre-ch14.18 Day 10 (Course 4 only): Post ch14.18 End of Treatment: Within 2 weeks post isotretinoin
Time Frame: PK samples obtained during Courses 1 and 3: Days 0, 3, 4, 5, 6, 7, 9, 10, 11, 14, 15, 16, 17; PK samples obtained during Courses 2 and 4: Days 0, 7, 10; End of Treatment
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Groups:
- UTC ch14.18: United Therapeutics Manufactured ch14.18
- NCI ch14.18: NCI Manufactured ch14.18
Arm/Group | UTC ch14.18 | NCI ch14.18
Number analyzed (Participants) | 27 | 27
mcg*hr/mL | 518 (418) | 470 (376)

2. Primary Outcome: Peak Plasma Concentration (Cmax)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | UTC ch14.18 | NCI ch14.18
Number analyzed (Participants) | 27 | 27
ng/mL | 6468 (719) | 6689 (853)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were reported at the time of informed consent through 30 days after the last dose of study therapy.
Arm/Group | UTC ch14.18 | NCI ch14.18
Serious Adverse Events (participants affected / at risk) | 17/27 | 12/27
Other Adverse Events (participants affected / at risk) | 27/27 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UTC ch14.18 (N=27) | NCI ch14.18 (N=27)
Device Related Infection (Infections and infestations) | 3 (3) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Alpha Hemolytic Stretococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (7) | 3 (7)
Disease Progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Serum Sickness (Immune system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Mydriasis (Eye disorders) | 1 (1) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Herpes Simplex (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Capillary Leak Syndrome (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UTC ch14.18 (N=27) | NCI ch14.18 (N=27)
Pyrexia (General disorders) | 27 (71) | 27 (64)
Pain (General disorders) | 16 (28) | 12 (22)
Platelet Count Decreased (Investigations) | 12 (18) | 12 (17)
Alanine Aminotransferase Increased (Investigations) | 18 (27) | 9 (15)
Neutrophil Count Decreased (Investigations) | 11 (19) | 9 (11)
Lymphocyte Count Decreased (Investigations) | 2 (3) | 4 (6)
White Blood Cell Count Decreased (Investigations) | 6 (8) | 8 (12)
Aspartate Aminotransferase Increased (Investigations) | 14 (27) | 14 (27)
Urine Output Decreased (Investigations) | 5 (11) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 25 (65) | 23 (55)
Hyponatremia (Metabolism and nutrition disorders) | 21 (48) | 20 (43)
Hypocalcemia (Metabolism and nutrition disorders) | 15 (30) | 15 (26)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (15) | 8 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 (60) | 26 (59)
Device Related Infection (Infections and infestations) | 4 (5) | 2 (2)
Gastroenteritis Viral (Infections and infestations) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 15 (22) | 13 (15)
Abdominal Pain (Gastrointestinal disorders) | 13 (22) | 11 (21)
Constipation (Gastrointestinal disorders) | 4 (7) | 3 (4)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 (14) | 11 (18)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
Hypotension (Vascular disorders) | 12 (18) | 9 (13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (21) | 14 (18)
Diarrhea (Gastrointestinal disorders) | 10 (13) | 13 (17)
Vomiting (Gastrointestinal disorders) | 10 (11) | 12 (21)
Nausea (Gastrointestinal disorders) | 9 (11) | 6 (10)
Cheilitis (Gastrointestinal disorders) | 1 (2) | 3 (3)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lip Swelling (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oropharyngeal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Face Odema (General disorders) | 10 (13) | 8 (9)
Fatigue (General disorders) | 5 (6) | 5 (10)
Malaise (General disorders) | 3 (5) | 3 (5)
Chills (General disorders) | 3 (3) | 2 (2)
Edema (General disorders) | 3 (4) | 3 (4)
Edema Peripheral (General disorders) | 4 (5) | 3 (3)
Injection Site Reaction (General disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 2 (2) | 1 (1)
Generalized Edema (General disorders) | 2 (2) | 0 (0)
Localized Edema (General disorders) | 1 (1) | 2 (2)
Blood Creatinine Increased (Investigations) | 3 (8) | 6 (6)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (4) | 5 (5)
Blood Bilirubin Increased (Investigations) | 6 (8) | 3 (6)
International Normalized Ratio Increased (Investigations) | 4 (6) | 3 (4)
Weight Decreased (Investigations) | 2 (2) | 3 (3)
Weight Increased (Investigations) | 3 (5) | 4 (5)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 3 (4) | 3 (5)
Electrocardiogram QT Prolonged (Investigations) | 2 (2) | 1 (1)
Blood Chloride Increased (Investigations) | 1 (2) | 2 (3)
Blood Triglycerides Increased (Investigations) | 2 (2) | 0 (0)
Eosinophil Count Increased (Investigations) | 2 (3) | 2 (3)
Gamma-Glutamyltransferase Increased (Investigations) | 2 (2) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 12 (14) | 10 (10)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (9) | 7 (8)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (8) | 4 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (5) | 8 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (18) | 7 (15)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 4 (7)
Fluid Retention (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 7 (10) | 7 (7)
Urticaria (Skin and subcutaneous tissue disorders) | 8 (9) | 6 (10)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 13 (21)
Rhinorrea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Capillary Leak Syndrome (Vascular disorders) | 6 (10) | 6 (9)
Hypertension (Vascular disorders) | 7 (15) | 7 (17)
Flushing (Vascular disorders) | 2 (2) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (5) | 1 (1)
Tachycardia (Cardiac disorders) | 11 (18) | 10 (15)
Sinus Tachycardia (Cardiac disorders) | 7 (14) | 7 (13)
Clostridium Difficile Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 7 (7) | 4 (7)
Hematuria (Renal and urinary disorders) | 2 (3) | 4 (5)
Proteinuria (Renal and urinary disorders) | 3 (5) | 5 (10)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 5 (8) | 4 (9)
Agitation (Psychiatric disorders) | 4 (7) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (4)
Abnormal Behavior (Psychiatric disorders) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 2 (2)
Periorbital Edema (Eye disorders) | 4 (4) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 2 (2)
Vision Blurred (Eye disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 1 (1)
Lethargy (Nervous system disorders) | 1 (2) | 2 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 3 (4) | 2 (3)
Hypoalbuminemia (Hepatobiliary disorders) | 3 (60) | 1 (59)
Hypersensitivity (Immune system disorders) | 2 (3) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed, except as provided below. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.